CLINICAL TRIAL: NCT04424953
Title: A Randomised Controlled Trial to Compare McGrath Videolaryngoscope Against Direct Laryngoscope for Endotracheal Intubation When Powered Air Purifying Respirator is Worn During the Current Coronavirus Disease 2019 Pandemic
Brief Title: To Compare Videolaryngoscope Against Direct Laryngoscope for Intubation When Powered Air Purifying Respirator is Worn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/2329
Record Dates: First submitted 2020-06-01; First posted 2020-06-11 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus Infection; Ventilatory Failure; Anesthesia Intubation Complication
Keywords: Intubation; Direct laryngoscope; Video laryngoscope; Personal protective equipment; Powered Air Purifying Respirator; Coronavirus Disease 2019
MeSH Terms: conditions — Coronavirus Infections; Hypoventilation; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Prior to a consented patient turning up for his/her operation, randomization will be done to determine who from the selected group of anesthetists will be doing the intubation. The randomly selected anesthetist will wear the PAPR and intubate the patient using either a DL or McGrath VL that he/she is randomized to.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients who have consented for the operation will not know which laryngoscope (either McGrath videolaryngoscope or direct laryngoscope) was used for their intubation. The outcomes assessor will not know which group the patients and the anesthetists are in when analysing the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- McGrath videolaryngoscope (Active Comparator): Anesthetists randomized to this group will intubate patients using the McGrath videolaryngoscope
  Interventions: Device: McGrath videolaryngoscope
- Direct laryngoscope (Active Comparator): Anesthetists randomized to this group will intubate patients using the direct laryngoscope
  Interventions: Device: Direct laryngoscope

INTERVENTIONS:
Device: McGrath videolaryngoscope — A brand of a commonly-used videolaryngoscope which has a camera at the end of the laryngoscope to visualize the vocal cords
  Arms: McGrath videolaryngoscope
Device: Direct laryngoscope — Classic direct laryngoscope that depends on visualization of the vocal cords by the operator
  Arms: Direct laryngoscope

SUMMARY:
Various guidelines for endotracheal intubation (insertion of breathing tube for mechanical ventilation) of Coronavirus Disease 2019 (COVID-19) patients recommend the use of videolaryngoscope (medical device used for intubation that has a camera to visualize the vocal cords between which the breathing tube will pass) over direct laryngoscope (conventionally-used medical device for intubation that depends on anesthetist's direct visualization of vocal cords). The reasons for this recommendation are to maximize the distance between the medical personnel and the patient's face during intubation to decrease the risk of viral particles transmission and to improve intubation success.

For patients infected with COVID-19, Powered Air Purifying Respirator (PAPR) is recommended as an alternative to N95 masks during aerosol-generating procedures such as intubation because N95 masks may not fully protect medical personnel from viral transmission during intubation.

There is no evidence to suggest that videolaryngoscope (VL) is superior to direct laryngoscope (DL) for intubation when PAPR is donned.

The purpose of this study is to determine if McGrath VL is superior to DL for intubation when the anesthetist is wearing a PAPR. The investigators' hypothesis is that McGrath VL will decrease the time to intubation by 20 seconds and more compared to DL when PAPR is donned. The investigators also hope to learn if there is any difference in the difficulties encountered between the use of VL and DL.

DETAILED DESCRIPTION:
Background:

17% of patients with Coronavirus Disease 2019 (COVID-19) may require endotracheal intubation for mechanical ventilation due to respiratory failure.

Various guidelines for endotracheal intubation of COVID-19 patients recommend the use of videolaryngoscope (VL) over direct laryngoscope (DL). The reasons for this recommendation are to firstly, maximize the distance between the medical personnel and the patient's face during intubation in order to decrease the risk of viral particles transmission and secondly, to improve intubation success.

There is a lack of evidence to show that VL can decrease the risk of contact with aerosol generated during intubation. Matthew T.V. Chan et al have shown that aerosol may be generated up to 45cm away from the patient's face during intubation. In the investigators' own trial run of an experimental set-up to study the difference in intubation between VL and DL when PAPR is worn, the investigators found that it is not possible to maintain a distance of at least 45cm during the intubation process because of the need to visualize the entry of the laryngoscope blade into the patient's mouth in order to prevent injury to the oral structures. The investigators' study is congruent with a recent study that reports the mean distance from the patient's mouth to anesthetist's mouth was 35.6cm using VL and 16.4cm using DL.

In routine intubations, VL is recommended over DL for endotracheal intubation as it may provide a higher success and faster speed of intubation compared to DL. For patients infected with COVID-19, PAPR is recommended as an alternative to N95 masks during aerosol-generating procedures such as intubation because N95 masks may not fully protect medical personnel from viral transmission during intubation. There is currently no evidence to suggest that VL is superior to DL for intubation when PAPR is donned.

Proposed Study Design:

This study will be a randomized controlled trial. Informed consent to take part in the study will be taken from patients who are planned for elective surgery requiring endotracheal intubation and also from a group of anesthetists in the department.

Prior to a consented patient turning up for the operation, randomization will be done to determine who from the selected group of anesthetists will be doing the intubation. The randomly selected anesthetist will wear the PAPR and intubate the patient using either a DL or McGrath VL that the anesthetist is randomized to.

Hypothesis and Objectives:

The hypothesis is that McGrath VL will decrease the time to intubation (TTI) by 20 seconds and more compared to DL when PAPR is donned. The investigators will also study the secondary outcomes between McGrath VL and DL which are first attempt success percentage, use of adjuncts, success or failure at intubation using initial laryngoscope that the anesthetists is randomized to, intubation difficulty scale (IDS), closest distance from patient's mouth to anesthetist's mouth during intubation, adverse events and inability to intubate despite all efforts by the anesthetist.

Sample size calculation:

The primary outcome of this study is the difference in time to complete intubation between DL and VL with hooded PAPR. In a previous study reported by Dong et al in 2013, 21 the median (IQR) time to complete tracheal intubation with suited VL was 18.2 (22.1 - 15.1 = 7.0) seconds, whereas that for suited DL was 26.4 (35.2 - 23.1 = 12.1) seconds.

For a normal distribution, the IQR which covers the middle 50% of the whole distribution is approximately equal to mean +/- 0.6 standard deviation (SD), or equivalently 1.2 SD. If time to complete intubation is normally distributed, the SD for suited VL and suited DL are approximately 5.8 and 10.1 seconds, respectively. To be conservative in calculating the sample size, the larger SD of 10.1 seconds for suited DL is used. Moreover, the distribution of time to complete intubation is unlikely normal but skewed, an inflated SD is assumed to compensate for the violation of normal distribution. Hence, a SD of 18 seconds is used.

The minimal clinically important difference (MCID) for time to complete intubation in comparing different laryngoscopes is not defined in the literature. MCIDs ranging between 10 and 20 seconds to compare intubation times using different laryngoscopes are commonly used, in this study a difference of 20 seconds is assumed. Therefore, to detect a difference of at least 20 seconds between the suited DL and suited VL groups, targeting a power of 80% and a 2-sided type I error of 5%, a sample size of 14 patients is required for each group (that is a total of 28 patients for the study).

The investigators will attempt to recruit 50 patients at the Pre-operative Evaluation Clinic (PEC) to account for a possible drop-out rate of 40% (either from patient refusal to take part in the study on the day of operation or from other unforeseen reasons why earlier-recruited patients will not be taking part in the study).

The investigators will recruit 10 anesthetists from the Division to increase the chance that the randomly selected anesthetist is available on the day of operation for a patient who has consented for the study.

Statistical analysis:

Data will be analyzed with an intention-to-treat analysis. To study the difference in TTI between McGrath VL and DL, the investigators will compare the mean or median time of for intubation with McGrath VL against DL using Mann-Whitney U test or Independent Samples T-test depending on the normality of the distribution.

To study the difference in the first-attempt success rate, use of adjuncts at first attempt, use of adjuncts at subsequent attempts, success or failure at intubation using initial laryngoscope randomized to, adverse events (oxygen desaturation to less than 88%, oro-dental injuries) and inability to intubate despite all measures between McGrath VL and DL, Chi-square test will be used. The investigators will compare the mean or median IDS for McGrath VL against that for DL and the mean or median of the closest distance between the patient's mouth and the anesthetist's mouth during intubation for McGrath VL against that for DL using Mann-Whitney U test or Independent Samples T-test depending on the normality of the distribution.

Quality assurance plan:

All data will be monitored and reviewed by the PI or Co-investigators. Training will be given to the clinical research coordinator for data extraction and entry to the case report forms for analysis will be verified by a second person from the study team. Records for all participants, including case report forms, all source documentation (containing evidence to study eligibility, history and physical findings, laboratory data, results of consultations, etc.) as well as Centralized Institutional Review Board (CIRB) records and other regulatory documentation will be retained by the PI and be accessible for inspection and copying by authorized authorities. The research data will be kept in the secure location within the departmental office for 7 years before being destroyed.

Safety monitoring:

Serious adverse event (SAE) in relation to human biomedical research, means any untoward medical occurrence as a result of any human biomedical research which:

* results in or contributes to death
* is life-threatening
* requires in-patient hospitalization or prolongation of existing hospitalization
* results in or contributes to persistent or significant disability/incapacity or
* results in or contributes to a congenital anomaly/birth defect
* results in such other events as may be prescribed Adverse event (AE) in relation to human biomedical research means any untoward medical occurrence as a result of any human biomedical research which is NOT serious. Adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease possibly/ probably/ definitely associated with the participant in the human biomedical research.

Only related SAEs (definitely/ probably/ possibly) will be reported to CIRB. Related means there is a reasonable possibility that the event may have been caused by participation in the research.

The investigator is responsible for informing CIRB after first knowledge that the case qualifies for reporting. Follow-up information will be actively sought and submitted as it becomes available.

Related AEs will not be reported to CIRB. However, the investigator is responsible to keep record of such AEs cases at the Study Site File.

Safety analyses and interim analyses will be done after 14 patients have completed the study to determine the incidence of adverse events. If there are more than 3 patients with adverse events, the investigators will review the safety of the study and decide if there is need to improve on the study design or terminate the study prematurely.

ELIGIBILITY:
Patients who attend the Pre-operative Evaluation Clinic (PEC) in Singapore General Hospital (SGH) for pre-anesthesia assessment will be screened by a study team member for recruitment if they meet the inclusion criteria.

Patients will be undergoing routine pre-anesthesia assessment (including review of medical conditions and airway anatomy) by the anesthetists in the PEC prior to their planned elective surgeries. During their routine pre-anesthesia assessment, they will also be assessed by a study team member to confirm if they meet the eligibility criteria. If they are eligible for enrollment, a qualified practitioner will take informed consent.

We will also recruit 10 anesthetists from the Division to perform the intubations. The 10 anaesthetists will have to self-report experience in both the use of McGrath videolaryngoscope (VL) and direct laryngoscope (DL) for intubation (at least 20 successful intubations with McGrath VL or DL).

Inclusion Criteria for patients:

* 21 years old and above
* Not pregnant
* ASA physical status I, II and III
* BMI less than 35kg/m2
* Elective surgical operations requiring general anesthesia and endotracheal intubation
* Able to give own informed consent
* No features of difficult airway which has to consist all of the following:
* Class I and II on the modified Mallampati classification
* Thyromental distance of 6.5cm and above
* Mouth opening of 3.5cm and above
* Sterno-mental distance of 12.5cm and above

Inclusion Criteria for Anesthetists:

* Qualified anesthetists (associate consultants and above)
* Experience with both the use of McGrath VL and DL for intubation (at least 20 successful intubations using McGrath VL)
* Willing to perform intubation with PAPR donned and using either the McGrath VL or DL

Exclusion Criteria for patients:

* Below 21 years old
* Pregnancy
* ASA status IV and above
* Poorly-controlled cardiorespiratory conditions (such as poorly-controlled asthma with Asthma Control Test ≤ 19, chronic obstructive pulmonary disease GOLD 2 and above, exertional angina, coronary artery disease with active symptoms, heart failure with New York Heart Association Class III and above)
* Body Mass Index ≥ 35 kg/m2
* Emergency operation
* Unable to give own consent
* Any feature of difficult airway which is
* Class III and IV on the Modified Mallampati Classification
* Thyromental distance less than 6.5cm
* Mouth opening less than 3.5cm
* Sterno-mental distance less than 12.5cm
* History of difficult intubation
* Unstable cervical spine

Exclusion criteria for anesthetists:

* Non-specialist anesthetist
* Inexperience with both the use of McGrath VL and DL for intubation (less than 20 successful intubations using McGrath VL)
* Unwilling to perform intubation with PAPR donned using either the McGrath VL or DL

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Time to intubation for McGrath videolaryngoscope versus direct laryngoscope | During the intubation process
  The time to intubation starts from the time the anesthetist takes over the laryngoscope till the first appearance of consecutive capnography tracings. The time to intubation will be assessed via a retrospective playback of the video-recording of the intubation process. Compares the time to intubation for McGrath videolaryngoscope against direct laryngoscope.

SECONDARY OUTCOMES:
Incidence of success at first intubation attempt with McGrath videolaryngoscope versus direct laryngoscope | During the intubation process
  Compares the incidence of success at first intubation attempt using McGrath videolaryngoscope against direct laryngoscope. To be assessed via a retrospective playback of the video-recording of the intubation process.
Incidence of the use of adjuncts at first attempt with McGrath videolaryngoscope versus direct laryngoscope | During the intubation process
  Compares the incidence of the use of adjuncts (bougie, stylet, external laryngeal pressure, hyper-angulated blades) at first attempt with McGrath videolaryngoscope against direct laryngoscope. To be assessed via a retrospective playback of the video-recording of the intubation process
Incidence of the use of adjuncts at subsequent attempts with McGrath videolaryngoscope versus direct laryngoscope | During the intubation process
  Compares the incidence of the use of adjuncts (bougie, stylet, external laryngeal pressure, hyper-angulated blades) at subsequent attempts (after first attempt) with McGrath videolaryngoscope against direct laryngoscope. To be assessed via a retrospective playback of the video-recording of the intubation process
Incidence of success and failure at intubation using initial laryngoscope | During the intubation process
  Compares the incidence of success and failure at intubation using the initial laryngoscope that the anesthetist is randomised to. To be assessed via a retrospective playback of the video-recording of the intubation process.
Intubation Difficulty Scale with McGrath videolaryngoscope versus direct laryngoscope | During the intubation process
  Compares the Intubation Difficulty Scale between using McGrath videolaryngoscope and direct laryngoscope for intubation. The scale is the sum of score from 7 variables. Ranges from 0 ("ideal" intubation, that is one performed without effort, on the first attempt, practiced by one operator, using one technique, full visualization of laryngeal aperture and vocal cords abducted) to infinity (impossible intubation). The higher the scale, the more difficulty the intubation process. To be assessed via a retrospective playback of the video-recording of the intubation process and also by interviewing the anesthetist who carried out the intubation.
Incidence of oxygen desaturation to less than 88% and oro-dental injuries with McGrath videolaryngoscope versus direct laryngoscope. | During the intubation process.
  Compares the incidence of oxygen desaturation to less than 88% and oro-dental injuries between the McGrath videolaryngoscope and direct laryngoscope. To be assessed during the playback of the video-recording of the intubation process and by interviewing the anesthetist.
Incidence of inability to intubate despite all efforts by the anesthetist with McGrath videolaryngoscope versus direct laryngoscope | During the intubation process
  Compares the incidence of inability to intubate despite all efforts by the anesthetist between the McGrath videolaryngoscope and the direct laryngoscope. To be assessed during the playback of the video-recording of the intubation process.
Closest distance from the patient's mouth to the anaesthetist's mouth during intubation | During the intubation process
  Compares the closest distance from the patient's mouth to the anaesthetist's mouth during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Qing Yuan Goh, M.Med (Anes), Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Brewster DJ, Chrimes N, Do TB, Fraser K, Groombridge CJ, Higgs A, Humar MJ, Leeuwenburg TJ, McGloughlin S, Newman FG, Nickson CP, Rehak A, Vokes D, Gatward JJ. Consensus statement: Safe Airway Society principles of airway management and tracheal intubation specific to the COVID-19 adult patient group. Med J Aust. 2020 Jun;212(10):472-481. doi: 10.5694/mja2.50598. Epub 2020 May 1. PMID 32356900
- [Result] Wax RS, Christian MD. Practical recommendations for critical care and anesthesiology teams caring for novel coronavirus (2019-nCoV) patients. Can J Anaesth. 2020 May;67(5):568-576. doi: 10.1007/s12630-020-01591-x. Epub 2020 Feb 12. PMID 32052373
- [Result] Zuo MZ, Huang YG, Ma WH, Xue ZG, Zhang JQ, Gong YH, Che L; Chinese Society of Anesthesiology Task Force on Airway Management; Airway Management Chinese Society of Anesthesiology Task Force on. Expert Recommendations for Tracheal Intubation in Critically ill Patients with Noval Coronavirus Disease 2019. Chin Med Sci J. 2020 Feb 27;35(2):105-9. doi: 10.24920/003724. Online ahead of print. PMID 32102726
- [Result] Cook TM, El-Boghdadly K, McGuire B, McNarry AF, Patel A, Higgs A. Consensus guidelines for managing the airway in patients with COVID-19: Guidelines from the Difficult Airway Society, the Association of Anaesthetists the Intensive Care Society, the Faculty of Intensive Care Medicine and the Royal College of Anaesthetists. Anaesthesia. 2020 Jun;75(6):785-799. doi: 10.1111/anae.15054. Epub 2020 Apr 1. PMID 32221970
- [Result] Chan MT, Chow BK, Chu L, Hui DS. Mask ventilation and dispersion of exhaled air. Am J Respir Crit Care Med. 2013 Apr 1;187(7):e12-4. doi: 10.1164/rccm.201201-0137im. No abstract available. PMID 23540885
- [Result] Hall D, Steel A, Heij R, Eley A, Young P. Videolaryngoscopy increases 'mouth-to-mouth' distance compared with direct laryngoscopy. Anaesthesia. 2020 Jun;75(6):822-823. doi: 10.1111/anae.15047. Epub 2020 Mar 29. No abstract available. PMID 32221979
- [Result] Lewis SR, Butler AR, Parker J, Cook TM, Smith AF. Videolaryngoscopy versus direct laryngoscopy for adult patients requiring tracheal intubation. Cochrane Database Syst Rev. 2016 Nov 15;11(11):CD011136. doi: 10.1002/14651858.CD011136.pub2. PMID 27844477
- [Result] Scales DC, Green K, Chan AK, Poutanen SM, Foster D, Nowak K, Raboud JM, Saskin R, Lapinsky SE, Stewart TE. Illness in intensive care staff after brief exposure to severe acute respiratory syndrome. Emerg Infect Dis. 2003 Oct;9(10):1205-10. doi: 10.3201/eid0910.030525. No abstract available. PMID 14609453
- [Result] Loeb M, McGeer A, Henry B, Ofner M, Rose D, Hlywka T, Levie J, McQueen J, Smith S, Moss L, Smith A, Green K, Walter SD. SARS among critical care nurses, Toronto. Emerg Infect Dis. 2004 Feb;10(2):251-5. doi: 10.3201/eid1002.030838. PMID 15030692
- [Result] Nouruzi-Sedeh P, Schumann M, Groeben H. Laryngoscopy via Macintosh blade versus GlideScope: success rate and time for endotracheal intubation in untrained medical personnel. Anesthesiology. 2009 Jan;110(1):32-7. doi: 10.1097/ALN.0b013e318190b6a7. PMID 19104167
- [Result] Altun D, Ali A, Camci E, Ozonur A, Seyhan TO. Haemodynamic Response to Four Different Laryngoscopes. Turk J Anaesthesiol Reanim. 2018 Dec;46(6):434-440. doi: 10.5152/TJAR.2018.59265. Epub 2018 Sep 6. PMID 30505605
- [Result] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Result] Roth D, Pace NL, Lee A, Hovhannisyan K, Warenits AM, Arrich J, Herkner H. Bedside tests for predicting difficult airways: an abridged Cochrane diagnostic test accuracy systematic review. Anaesthesia. 2019 Jul;74(7):915-928. doi: 10.1111/anae.14608. Epub 2019 Mar 6. PMID 30843190
- [Result] Cormack RS, Lehane J. Difficult tracheal intubation in obstetrics. Anaesthesia. 1984 Nov;39(11):1105-11. PMID 6507827
- [Result] Greenland KB, Tsui D, Goodyear P, Irwin MG. Personal protection equipment for biological hazards: does it affect tracheal intubation performance? Resuscitation. 2007 Jul;74(1):119-26. doi: 10.1016/j.resuscitation.2006.11.011. Epub 2007 Mar 13. PMID 17353076
- [Result] Shin DH, Choi PC, Na JU, Cho JH, Han SK. Utility of the Pentax-AWS in performing tracheal intubation while wearing chemical, biological, radiation and nuclear personal protective equipment: a randomised crossover trial using a manikin. Emerg Med J. 2013 Jul;30(7):527-31. doi: 10.1136/emermed-2012-201463. PMID 23765764
- See also: Liana Zucco, Nadav Levy, Desire Ketchandji, Mike Aziz, S. K. R. Anesthesia Patient Safety Foundation - Perioperative Considerations for the 2019 Novel Coronavirus (COVID-19) — https://www.apsf.org/news-updates/perioperative-considerations-for-the-2019-novel-coronavirus-covid-19/
- See also: Australian Society of Anaesthetists. COVID-19 Updates. — https://asa.org.au/covid-19-updates/